CLINICAL TRIAL: NCT02503098
Title: Optimizing a Smartphone Application for Individuals With Eating Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Recovery Record Research (Industry)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RRR-023
Record Dates: First submitted 2015-07-15; First posted 2015-07-20 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Eating Disorders; Binge Eating Disorder; Bulimia Nervosa
Keywords: Eating Disorders; Cognitive Behavioral Therapy; Mobile Phone; Smartphone; App; Binge Eating Disorder; Bulimia Nervosa; Signal Detection Analysis
MeSH Terms: conditions — Feeding and Eating Disorders; Binge-Eating Disorder; Bulimia Nervosa; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Recovery Record adaptive smartphone application (RR-A) (Experimental): Participants will have access to all Recovery Record standard functions and will additionally receive tailored, algorithm-generated content targeting cognitive distortions.
  Interventions: Behavioral: Recovery Record adaptive smartphone application
- Recovery Record standard smartphone application (RR-S) (Active Comparator): Participants will have access to all Recovery Record standard functions, including meal monitoring, motivational enhancement, social support, and coping skill strategies.
  Interventions: Behavioral: Recovery Record standard smartphone application

INTERVENTIONS:
Behavioral: Recovery Record adaptive smartphone application
  Arms: Recovery Record adaptive smartphone application (RR-A)
Behavioral: Recovery Record standard smartphone application
  Arms: Recovery Record standard smartphone application (RR-S)

SUMMARY:
This study will augment an existing mobile application for individuals with eating disorders by developing adaptive, tailored content targeting remediation of cognitive distortions. The adaptive application will be deployed and assessed for efficacy relative to the standard product in a randomized controlled trial.

DETAILED DESCRIPTION:
Eating Disorders (ED) are common and serious psychological disorders. Anorexia Nervosa (AN) has a prevalence estimated at between 0.48% and 0.70% among young females. Bulimia Nervosa (BN) is a serious mental health problem, with a prevalence of between 1-2% of young women while clinically significant bulimic behaviors occur in an additional 2-3%. There are significant barriers to access of evidence-based treatments and current models of individual psychotherapy will likely never meet the enormous need for psychological services for ED. Unfortunately, even with treatment, rates of recovery are modest with the best performing treatments achieving remission in only about 50% of cases while relapse rates are high, especially if the ED becomes chronic. It is widely acknowledged that a major shift in intervention practice is needed and that smartphone apps will almost certainly play a role due to their reach and breadth of functionality.

As the first commercially available smartphone app for EDs, Recovery Record (RR) has established wide reach and user acceptability. The app provides users with meal and ED symptom self-monitoring and coping skill strategies in an evidence-based CBT format. Preliminary pilot data suggest that for a proportion of RR users, using RR is associated with clinically significant symptom reduction. However, a limitation of the current app is that it is a "one-size-fits-all" product that does not account for the heterogeneity of ED symptoms. Genetic, personality and neurocognitive data support distinct clusters of ED presentations that also differ according to response to treatment, course and outcome. Pilot data confirm that clinical response to RR is not homogenous across groups and that extent of cognitive distortions is the most potent factor to predict outcome. There is considerable opportunity to increase RR's effectiveness across a range of ED symptoms and behaviors by creating adaptive and tailored content focused on remediation of cognitive distortions.

During Phase 1 of this study screening algorithm will be validated against an unseen, prospective test dataset of approximately 2,000 users. All candidate predictor variables will be entered into a Signal Detection Analysis to confirm the sensitivity and specificity of the screen. Informed by the resultant algorithms, adaptive content will be developed that targets ED-specific cognitive distortions. To evaluate acceptability, adapted content will be piloted with approximately 200 individuals for a period of one month. Participant feedback and utilization data will inform content acceptability and feasibility. By the end of the first phase tailored content that is acceptable to individuals with specific symptom presentations will be developed.

Phase 2 will focus on an evaluation of whether an adaptive app offering tailored content addressing eating related cognitive distortions in a stepped way can outperform the current standard app. The adaptive content will be integrated into a new, dynamic version of the app (RR-A) that will then be evaluated against the current app (RR-S). Approximately 5,000 registered users of RR will be randomized to receive either RR augmented with targeted content (RR-A), or RR in its current standard format (RR-S) over a two-month period. Outcome data will be measured at baseline, one month, end of treatment, and at six-month follow-up. At the end of the study period it is predicted that the resultant evidence-based product will have demonstrated ability to bring about clinically significant reduction in symptoms in more users than the current app, and thus will have potential to make a substantial public health impact.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for clinically significant symptoms of eating disorder using self-report measures
* Has an Android or iPhone and is willing to use phone for the study
* Is able to speak and read English
* Lives within the United States of America
* Is at least 16 years of age

Exclusion Criteria:

* Has visual, hearing, voice, or motor impairment that would prevent completion of study and treatment procedures
* Has any psychiatric condition for which participation in a clinical trial of psychotherapy may be either inappropriate or dangerous (e.g., psychotic disorders, bipolar disorders, severe post traumatic stress disorder, etc.).
* Exhibits severe suicidality, including ideation, plan, and intent.
* Currently receiving weekly psychotherapy or planning to receive weekly psychotherapy for eating disorder during the 12 weeks of the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3340 (Actual)
Dates: Start 2016-11-23 (Actual); Primary Completion 2018-07-13 (Actual); Study Completion 2018-09-13 (Actual)

PRIMARY OUTCOMES:
Changes in Eating Disorder Severity | Measured at the start of treatment (baseline), week 4, week 8 and 6 months follow-up
  Self-reported eating disorder symptom severity. To measure changes in eating disorder severity over time, the Eating Disorder Evaluation Questionnaire (EDE-Q) will be used.

SECONDARY OUTCOMES:
Binge eating and purging episode frequency | Measured at the start of treatment (baseline), week 4, week 8 and 6 months follow-up
  Self-reported disordered behavior frequency will be assessed via behaviors self-monitored in the application in addition to symptom frequency questions in the Eating Disorder Evaluation Questionnaire.
Changes in Clinical Impairment Severity | Measured at the start of treatment (baseline), week 4, week 8 and 6 months follow-up
  To measure changes in eating disorder related clinical impairment over time, the self-reported Clinical Impairment Assessment (CIA) will be used.
Participant Satisfaction | Participants will be followed for the duration of the 8-week trial
  Self-reported satisfaction
Adherence to the mobile application intervention | Measured from the start of application utilization (baseline) to 8-weeks
  Adherence will be measured via dichotomous outcome of drop-out (an individual will be considered a system drop-out if they fail to login to the app at all for a period of 14 consecutive days). Adherence will be assessed through application usage data.
Adherence to self-monitoring tasks | Measured from the start of application utilization (baseline) to 8-weeks
  Frequency of self-monitoring entries will be tracked automatically through the program server.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Recovery Record Research, San Francisco, California
  - Stanford University School of Medicine, Department of Psychiatry and Behavioral Sciences, Stanford, California

REFERENCES:
- [Derived] Tregarthen J, Paik Kim J, Sadeh-Sharvit S, Neri E, Welch H, Lock J. Comparing a Tailored Self-Help Mobile App With a Standard Self-Monitoring App for the Treatment of Eating Disorder Symptoms: Randomized Controlled Trial. JMIR Ment Health. 2019 Nov 21;6(11):e14972. doi: 10.2196/14972. PMID 31750837
- See also: Recovery Record smartphone application website — http://www.recoveryrecord.com